CLINICAL TRIAL: NCT04440839
Title: Implementation of Telemedicine for Patient With Lower Extremity Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1598596; 5K23HL143178-05 (NIH)
Record Dates: First submitted 2020-06-11; First posted 2020-06-22 (Actual); Results first posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Peripheral Arterial Disease; Peripheral Artery Disease; Peripheral Vascular Diseases; Diabetic Foot; Diabetic Foot Ulcer; Diabetic Foot Infection; Diabetic Peripheral Neuropathy
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases; Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Patients identified as having a lower extremity wound with peripheral artery disease or diabetes mellitus are offered a telemedicine consult. Patients are then followed for time to consultation, time to revascularization if needed, and time to wound healing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Telemedicine specialty consultation for patients
  Interventions: Other: Telemedicine specialty consultation
- Standard Care (No Intervention): Standard in person referral to a specialist

INTERVENTIONS:
Other: Telemedicine specialty consultation — Patients with lower extremity wounds due to peripheral artery disease and diabetes mellitus will undergo a specialty consultation with a provider through telemedicine
  Arms: Intervention

SUMMARY:
The objective of this study is to determine if patients with lower extremity wounds in rural communities who undergo specialty referral through telemedicine have expedited care compared to patients who are treated through standard in person referral.

DETAILED DESCRIPTION:
This is a clustered trial where patients identified as having lower extremity ulcers with peripheral artery disease and diabetes are given the option to be seen by specialty care providers through telemedicine vs. normal standard in person referral. The study is being conducted in rural areas where there are no in person vascular surgery providers. The aim of the study is to determine if patient activation affects likelihood to use telemedicine and if use of telemedicine can expedite speciality care.

ELIGIBILITY:
Inclusion Criteria:

* Patient with the diagnosis of a lower extremity ulcer that has been present for longer than 2 weeks
* Must be willing to complete the patient activation survey
* Must be willing to have the study personnel call them to check in on their status

Exclusion Criteria:

* Patients that do not have a telephone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Misty D Humphries, Principal Investigator — University of California, Davis
Locations (1):
- Misty D. Humphries, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from two clinical sites where wound care was provided. One site had access to revascularization services and the other did not.
Pre-assignment Details: All subjected had to have a wound on the foot.
Groups:
- Telemedicine: Participants received specialty wound care consultations through telemedicine.
- Standard Care: Participants received usual wound care at their clinic without telemedicine consultation.
Period: Overall Study
Arm/Group | Telemedicine | Standard Care
Started | 116 | 0
Completed | 113 | 0
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Population: Baseline demographic and clinical characteristics were collected for participants in both the Telemedicine and Standard Care arms.
Groups:
- Telemedicine: Telemedicine specialty consultation for patients These subjects were all >18 years old, of all races specifically with a focus on the native American population is the area of one clinic.
- Standard Care: Patent who received wound care without telemedicine
- Total: Total of all reporting groups
Arm/Group | Telemedicine | Standard Care | Total
Number analyzed (Participants) | 113 | 0 | 113
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 69 [61 to 77] |  | 69 [61 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 0 | 38
  Male | 75 | 0 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 0 | 20
  Not Hispanic or Latino | 91 | 0 | 91
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 5 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 12 | 0 | 12
  White | 73 | 0 | 73
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 19 | 0 | 19

OUTCOME MEASURES:

1. Primary Outcome: Specialty Consultation
Description: The time from the date the wound is identified to the date of specialist consultation, in days.
Time Frame: up to 365 days
Population: Due to COVID-19-related changes at the time the study was initiated, no subjects were enrolled in the standard car group.
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- Intervention: Telemedicine specialty consultation for patients These subjects were all >18 years old, of all races specifically with a focus on the native American population is the area of one clinic.
- Standard Care: Subjects who received wound care without a telemedicine visit
  NO subjects were enrolled in this group due to COVID restrictions and changes in subject participation
Arm/Group | Intervention | Standard Care
Number analyzed (Participants) | 113 | 0
days | 66 [33 to 139] |

2. Secondary Outcome: Revascularization
Description: The time from the date the wound is identified to the procedure to evaluation or improve blood flow for the index leg, in days.
Time Frame: up to 365 days
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- Standard Care: Subjects who had wound care without telemedicine consult
Arm/Group | Intervention | Standard Care
Number analyzed (Participants) | 113 | 0
days | 71 [16 to 245] |

3. Secondary Outcome: Wound Healing
Description: The time from when the wound is identified until the wound heals, in days.
Time Frame: up to 365 days
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Intervention | Standard Care
Number analyzed (Participants) | 113 | 0
days | 174 [76 to 402] |

4. Secondary Outcome: Amputation
Description: Major (above the ankle) or minor (toe/TMA) amputation of the index leg.
Time Frame: up to 365 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Standard Care
Number analyzed (Participants) | 113 | 0
Participants
  No amputation | 83 |
  minor amputation | 20 |
  Major amputation | 5 |
  Lost to follow up | 5 |

ADVERSE EVENTS:
Time Frame: From enrollment until completion of follow-up at 6 months.
Description: Death and lost to follow up before healing was considered an adverse event
Groups:
- Standard Care: Subjects who had wound care without a telemedicine consultation
Arm/Group | Intervention | Standard Care
All-Cause Mortality (participants affected / at risk) | 3/113 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/113 | 0/0
Other Adverse Events (participants affected / at risk) | 0/113 | 0/0

LIMITATIONS AND CAVEATS:
A significant limitation was the absence of a comparator group for subjects at the most remote telemedicine clinic. However, we were able to enroll subjects and provide them with improved care in the intervention group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/39/NCT04440839/Prot_SAP_000.pdf